CLINICAL TRIAL: NCT05055193
Title: Outcome of Extremely Preterm Infants Who Received Systemic Postnatal Corticosteroid for Bronchopulmonary Dysplasia
Acronym: DEPRECOD
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2021_005
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm infants who received postnatal corticosteroid for bronchopulmonary dysplasia: Corticosteroids used are hydrocortisone (as first-line therapy) and betamethasone (in situations of particular severity)
  Interventions: Drug: Evaluation at 24 months corrected age: respiratory outcome, Neurodevelopmental outcome, Growth outcome
- Preterm infants who did not receive postnatal corticosteroid for bronchopulmonary dysplasia: No corticosteroids

INTERVENTIONS:
Drug: Evaluation at 24 months corrected age: respiratory outcome, Neurodevelopmental outcome, Growth outcome — Data concerning the 24 months corrected age outcomes were collected from the medical records of the ECL'AUR preterm infants follow-up network.
  Groups: Preterm infants who received postnatal corticosteroid for bronchopulmonary dysplasia

SUMMARY:
Bronchopulmonary dysplasia is a complication of prematurity. Postnatal corticosteroid is used to treat the inflammatory part of this pathology, in particular to wean premature infants from the ventilator at the end of the first month of life. However, this therapy remains controversial because it may induce suboptimal neurocognitive development. Parents of infants who receive postnatal corticosteroid should be provided with information about the risks. The objective of our work was to evaluate the respiratory, neurodevelopmental and growth outcomes at 24 months corrected age of extremely preterm infants who received postnatal corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* Extremely preterm infants less than 29 weeks' gestation
* Infants hospitalized for at least the first 30 days of life in the neonatology department of the Croix-Rousse Hospital in Lyon
* Infants born between January 1, 2013 and December 31, 2016

Exclusion Criteria:

* Infants with a congenital heart, lung or brain malformation
* Infants with a neuromuscular disease
* Infants with a genetic disorder
* Infants who died before the age of 24 months corrected age
* Infants lost to follow-up or with incomplete data at 24 months corrected age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extremely preterm infants less than 29 weeks' gestation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Composite primary outcome combining: - Respiratory evolution at 24 months corrected age - Neurodevelopmental evolution at 24 months corrected age - Growth evolution at 24 months corrected age | at 24 months corrected age
  * Respiratory evolution at 24 months corrected age: asthma, inhaled corticosteroid therapy, respiratory events, hospitalizations for respiratory events.
  * Neurodevelopmental evolution at 24 months corrected age: developmental quotient of the revised Brunet Lézine scale, visual and auditory anomalies, cerebral palsy.
  * Growth evolution at 24 months corrected age: weight, height and head circumference at 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civil de Lyon, Lyon, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Derived] Melan N, Pradat P, Godbert I, Pastor-Diez B, Basson E, Picaud JC. Neurodevelopment at 24 months corrected age in extremely preterm infants treated with dexamethasone alternatives during the late postnatal period: a cohort study. Eur J Pediatr. 2024 Feb;183(2):677-687. doi: 10.1007/s00431-023-05319-z. Epub 2023 Nov 13. PMID 37955745